CLINICAL TRIAL: NCT01471873
Title: Variability of Pentacam-derived Back Elevation Measurements in Keratoconus and Cross-linked Corneas
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Senior Lecturer of Ophthalmology, Democritus University of Thrace
Other Study IDs: 25/27-09-2011
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Keratoconus
Keywords: Posterior corneal surface elevation; Pentacam-Scheimpflung imaging; variability; progressive keratoconus; corneal cross-linking
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Keratoconus Group (KG): Keratoconus group (KG) included patients with progressive keratoconus.
- Collagen-Cross-linking group (CXLG): Collagen-Cross-linking group (CXLG) included keratoconus patients that had been treated with uneventful corneal collagen cross-linking (CXL) at least on year prior to their enrolment in the study.
  Interventions: Procedure: Corneal Collagen Cross-linking (CXL)

INTERVENTIONS:
Procedure: Corneal Collagen Cross-linking (CXL) — The same surgical procedure was applied to all CXLG patients that included:
  Instillation of proparacaine hydrochloride 0.5% drops for topical anaesthesia, application of a sponge saturated with 10% alcohol to the central cornea for 20-30 seconds and subsequent de-epithelialization by means of a hockey knife. Following de-epithelialization, a mixture of 0.1% riboflavin in 20% Dextran solution was instilled to the cornea for 30 minutes (2 drops every 2 minutes) prior to the irradiation. In details, an 8.0mm diameter of central cornea was irradiated for 30 minutes by UVA light with a wavelength of 370nm and an irradiance of 3mW/cm2.The UVA radiation source that was used is the UV-XTM (IROC AG, Zurich, Switzerland). Instillation of riboflavin drops (1 drop every 2 minutes) was continued during irradiation, as well.
  Groups: Collagen-Cross-linking group (CXLG)

SUMMARY:
Primary objective of this study was to assess the intrasession, intersession and interobserver variability of the Pentacam-derived posterior corneal elevation measurements in keratoconus eyes and eyes that underwent Corneal Collagen Cross-liknking (CxL) treatment due to progressive keratoconus.

DETAILED DESCRIPTION:
The Pentacam Classic (Oculus Optikgerate GmbH, Heidelberg, Germany, software version 1.14r04) was used for the sake of the study.Two study groups were formed: 1) Keratoconus group (KC) included patients with progressive keratoconus and 2) Collagen-Cross-linking group (CXL) included keratoconus patients that had been treated with uneventful CXL at least on year prior to their enrollment in the study.

Three consecutive scans were obtained by two experienced operators. The same procedure was repeated within two weeks for the assessment of intersession variability. In all cases acceptable maps had at least 10.0mm of corneal coverage.All back elevation points were codified in order to facilitate statistical processing of data. Further to single point analysis, three additional parameters were evaluated: a) zone 4 parameter (z4) which derived by the analysis of all points at the central 4.0mm diameter zone, b) zone 8 parameter (z8) which derived by the analysis of all points at the central 8.0mm diameter zone, and, c) highest elevation point parameter (HEP), which derived by the analysis of the highest elevation points for all participants. Reproducibility of measurements was evaluated by means of intraclass correlation coefficients (ICC). Three different ICC types were calculated: a) intrasession ICC for both operators (ICC1 & ICC2), b) interobserver ICC, and, c) intersession ICC. Moreover, Bland-Altman plots were used to evaluate the level of agreement between the two operators.

ELIGIBILITY:
Inclusion Criteria:

* Progressive keratoconus (Keratoconus group)
* Corneal collagen cross linking (CxL) treatment at least one year prior to enrollment (CxL group)

Exclusion Criteria:

* Glaucoma
* Suspicion of glaucoma
* history of herpetic keratitis
* corneal scarring
* severe eye dryness
* pregnancy or nursing
* current corneal infection
* underlying autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from the Cornea service of the EIT in a consecutive-if-eligible basis.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Variability of posterior corneal surface elevation measurements within and between sessions and within and between observers. | 2 weeks
  The Pentacam Classic (Oculus Optikgerate GmbH, Heidelberg, Germany, software version 1.14r04) was used for the sake of the study. Three consecutive scans were obtained by two experienced operators for the assessment of intrasession and interobserver variability. The same procedure was repeated within two weeks for the assessment of intersession variability.Bland-Altman plots were used to evaluate agreement between the 2 operators. The reproducibility of all measurements was evaluated by means of the intraclass correlation coefficient(ICC).

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute of Thrace (EIT), Alexandroupoli, Thrace, Greece

REFERENCES:
- [Result] Labiris G, Giarmoukakis A, Sideroudi H, Bougatsou P, Lazaridis I, Kozobolis VP. Variability in Scheimpflug image-derived posterior elevation measurements in keratoconus and collagen-crosslinked corneas. J Cataract Refract Surg. 2012 Sep;38(9):1616-25. doi: 10.1016/j.jcrs.2012.04.039. PMID 22906447